CLINICAL TRIAL: NCT06198218
Title: Effects of Activity Based Scapular Mobilization on Upper Limb Function in Children With Erbs Palsy
Brief Title: Effects of Scapular Mobilization on Upper Limb Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: REC/RCR&AHS/23/0756
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Erbs Palsy
Keywords: Erbs palsy; scapular mobilization; mallet score; codman exercises
MeSH Terms: conditions — Brachial Plexus Neuropathies

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will get separate treatment protocol as and possible efforts will be put to mask the both groups about their treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scapular mobilization (Experimental): This Experimental group will be treated with manual scapular mobilization in upward rotation and downward rotation, adduction and abduction of scapula. Sets of 10 repetitions were applied with a rest interval of 30 seconds between set for 20 minutes, activity based scapular mobilization(Codman pendulum exercises, scapular pushups, band wall apart ,wall ball circles and advance study wall pushups) along with conventional physical therapy program(heating,EMS,stretching for tight muscles , strengthening exercises and graduated active exercises) for 25 minutes
  Interventions: Other: Scapular mobilization
- Conventional physical therapy program (Active Comparator): This group will receive conventional physical therapy program including ( heating to improve circulation and release muscle tension ,EMS ,stretching for stiff muscle, weight bearing, strengthening exercises and graduated active exercises)for 20 minutes along with activity based scapular mobilization( Codman pendulum exercises, ban wall apart, wall ball circles, scapular pushups and advance study wall pushups)for 20 minutes with 5 minute resting interval.
  Interventions: Other: Conventional physical therapy program

INTERVENTIONS:
Other: Scapular mobilization — Group A: will be treated with manual scapular mobilization in upward rotation and downward rotation, adduction and abduction of scapula.Sets of 10 repetitions were applied with a rest interval of 30 seconds between set for 20 minutes, activity based scapular mobilization(Codman pendulum exercises, scapular pushups, band wall apart ,wall ball circles and advance study wall pushups) along with conventional physical therapy program(heating,EMS,stretching for tight muscles , strengthening exercises and graduated active exercises) for 25 min
  Other Names: Standard
  Arms: Scapular mobilization
Other: Conventional physical therapy program — Group B:will receive conventional physical therapy program including (heating to improve circulation and release muscle tension,EMS,stretching for stiff muscle,weight bearing, strengthening exercises & graduated active exercises)for 20 min along with activity based scapular mobilization (Codman pendulum exercises,band wall apart,wall ball circles, scapular pushups and advance study wall pushups)for 20 min with 5 min resting interval.
  Arms: Conventional physical therapy program

SUMMARY:
Erb's Palsy is a physical impairment resulting from an injury to the upper trunk of the brachial plexus and is associated with paralysis of the upper limb. When the neck is stretched up and move away from the wounded shoulder while the shoulder is pressed down, damage to the top nerves that make up the brachial plexus is more likely to damage .These injuries occur due to traumatic activities(vehicle accidents),difficult births(breeched presentation ,prolonged labor and high birth weight).This study proposes to analyze the effects of activity based scapular mobilization on upper limb functions in children who have been diagnosed with Erb's Palsy.

This will be a randomized control trial study. Data will be collected from 30 patients who will be randomly assigned to two groups of equal numbers experimental and control group each with 15. The participants of the experimental group will be treated with scapular mobilization ,activity based scapular mobilization(codman pendulum exercises,scapular pushups, band wall apart,wall ball circles and advance study wall pushups) along with conventional physical therapy program. Participants of control group is treated with activity based scapular mobilization and conventional physical therapy program. Patient evaluation will be made at the beginning and end of the treatment. Data will be analyzed through SPSS 25.

DETAILED DESCRIPTION:
Data will be collected from M.Islam teaching hospital Gujranwala and district health quarter Gujranwala .30 patients will be randomly assigned into two groups of equal numbers experimental and control group each with 15. Control group will receive conventional physical therapy program including ( heating to improve circulation and release muscle tension ,EMS ,stretching for stiff muscle, weight bearing, strengthening exercises and graduated active exercises)for 20 minutes along with activity based scapular mobilization( Codman pendulum exercises, ban wall apart, wall ball circles, scapular pushups and advance study wall pushups)for 20 minutes with 5 minute resting interval. Experimental group will be treated with manual scapular mobilization in upward rotation and downward rotation, adduction and abduction of scapula. Sets of 10 repetitions were applied with a rest interval of 30 seconds between set for 20 minutes, activity based scapular mobilization(Codman pendulum exercises, scapular pushups, band wall apart ,wall ball circles and advance study wall pushups) along with conventional physical therapy program(heating,EMS,stretching for tight muscles , strengthening exercises and graduated active exercises) for 25 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 6-9 years
* Diagnosed as obs. Erb's palsy
* Able to perform exercise
* Unilateral involvement of shoulder joint
* Unilateral active and passive movement of shoulder joint
* Both male and female involved
* Willing to participate

Exclusion Criteria:

* No history of surgery (arthroscopy, fixations)
* Any skin condition ( Allergies, infection)
* Local corticosteroids injections into the effected shoulder over last 3 months
* No present Fracture/ contractures
* Neurological disorders with muscle weakness in shoulder joint .

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
range of motion | 8 weeks
  A goniometer is a tool used to measure angles. It is an important tool for those studying anatomy, helping to measure the range of motion in joints. Goniometers are also used in physical therapy, engineering, and other fields.
functional capacity | 8 weeks
  Box-and-block tests are a type of physical evaluation used to measure an individuals lateral rotation. Angles are measured from video stills for abduction, hand to mouth and apparent supination and estimated for lateral rotation.

CONTACTS AND LOCATIONS:
Overall Officials: Amina Bibi, MS*, Principal Investigator — Riphah International Univeristy
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ho ES, Curtis CG, Clarke HM. The brachial plexus outcome measure: development, internal consistency, and construct validity. J Hand Ther. 2012 Oct-Dec;25(4):406-16; quiz 417. doi: 10.1016/j.jht.2012.05.002. Epub 2012 Jul 20. PMID 22818900